CLINICAL TRIAL: NCT02282241
Title: A Randomized Double-Blind Placebo-Controlled Study on the Use of Melatonin for the Prevention of Delirium
Brief Title: Melatonin for Delirium Prophylaxis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Project never began
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Peter Y Chan, Dr. Peter Chan, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H13-02843
Record Dates: First submitted 2014-10-30; First posted 2014-11-04 (Estimated); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Delirium
Keywords: Melatonin; Sleep; Delirium
MeSH Terms: conditions — Delirium | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients given once daily placebo (cellulose) orally in the evening, for 14 days.
  Interventions: Other: Placebo
- Melatonin (Experimental): Patients given once daily melatonin 1.5mg orally in the evening, for 14 days.
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin
  Arms: Melatonin
Other: Placebo
  Arms: Placebo

SUMMARY:
Delirium is a common complication of illness especially among the elderly with serious sequelae including increased mortality, morbidity and length of stay. This neuropsychiatric emergency has key features including acute onset, fluctuating level of consciousness, poor attention and cognitive deficits with a presentation which may include hallucinations and delusions.

A critical precipitating and maintaining feature of delirium is disrupted sleep. Melatonin is a widely available natural health product with evidence in normalizing circadian rhythms and sleep. There is also preliminary evidence that melatonin can be used to prevent the development of delirium in hospitalized patients. We hypothesize that daily administration of melatonin (1.5mg) in the evening, beginning at first admission to hospital and continuing for 14 days, will lead to decreased rates of delirium compared to placebo-treated comparison subjects.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or greater
* Admitted to hospital under the care of the hospitalist service or sub-acute medicine wards.

Exclusion Criteria:

* those who are suspected to be delirious at the time of their initial presentation;
* those who are already taking melatonin prior to admission;
* those who are not expected to live more than 48 hours;
* those suffering severe dementia (as indicated by a score of 6-7 on the Global Deterioration Scale adapted by Dr. Doug Drummond from Reisberg et al. (Reisberg 1982);
* those who are unable to reliably take oral medications;
* those presenting with an intracranial bleed, seizure or acute stroke;
* those with a known allergy or adverse reaction to the study compounds;
* those who cannot be evaluated initially because of depressed level of consciousness or inability to communicate;
* those anticipated to require surgery early in their hospitalization.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Delirium (Confusion Assessment Method) | Within 14 days
  Screening will be performed by a research assistant using the Confusion Assessment Method, and those with positive screening diagnosed by a study physician.

SECONDARY OUTCOMES:
Confusion (Confusion Assessment Method scores) | Within 14 days
  Confusion Assessment Method scores.
Mortality | Within 14 days
Use of restraints | Within 14 days
Code White (Violence) | Within 14 days

OTHER OUTCOMES:
Length of Stay | Within 6 months
Time to delirium | Within 14 days
Discharge Functional Status (Physiotherapist or Occupational therapist assessed) | Within 6 months
  Physiotherapist or Occupational therapist assessed
Discharge Disposition (Unchanged from pre-admission Home Home with supports Rehabilitation Assisted living) | Within 6 months
  Unchanged from pre-admission Home Home with supports Rehabilitation Assisted living
Sleep (Hours slept according to nursing records) | Within 14 days
  Hours slept according to nursing records

CONTACTS AND LOCATIONS:
Overall Officials: Peter KY Chan, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver Coastal Health, Vancouver, British Columbia, Canada